CLINICAL TRIAL: NCT00034190
Title: A Phase IIa Multicenter Evaluation of The Safety And Efficacy of Weekly Administration of S-8184 Paclitaxel Injectable Emulsion In Second Line Treatment of Patients With Stage III or IV Colorectal Adenocarcinoma
Brief Title: Safety and Efficacy of S-8184 in Second Line Treatment of Stage III or IV Colorectal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Monica S. Krieger, VP Regulatory Affairs, OncoGenex Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SON-8184-1066
Record Dates: First submitted 2002-04-23; First posted 2002-04-25 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Colorectal Adenocarcinoma

INTERVENTIONS:
Drug: S-8184 Paclitaxel Injectable Emulsion

SUMMARY:
Phase IIA, multicenter, dose escalation study evaluating the safety and efficacy of weekly S-8184 paclitaxel injectable emulsion in second line treatment of patients with stage III or IV colorectal adenocarcinoma.

DETAILED DESCRIPTION:
The goals of this study are to determine the objective response rate, to determine time to disease progression, duration of response, and survival, and to identify the maximum tolerated weekly dose and principal toxicities of S-8184 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

Histologic diagnosis of colorectal adenocarcinoma

Stage III or IV (Dukes's stage C or D)

One and only one prior cytotoxic chemotherapy regimen which must have included 5-FU

Adult (18 years of age or older) patients

Adequate hematologic function (ANC greater than 1500 cells/mm3 and platelets greater than 100,000/mm3)

Serum creatinine less than 2.0 mg/dL

Total bilirubin less than 1.5 mg/dL; SGOT and SGPT less than 3 times the upper limit of institutional normal values

ECOG performance status of 0 - 2

Bidimensional measurable disease

Patients who have signed an IRB / Ethics Committee approved informed consent

Life expectancy at least 12 weeks

Patient has fully recovered from any previous surgery (at least 4 weeks since major surgery)

Patient has a negative pregnancy test prior to study entry if premenopausal. (Patients of child bearing potential must use a medically effective form of contraception during the treatment.)

Exclusion Criteria:

Patients who have received any taxane-containing preparation including Taxol (paclitaxel) or Taxotere (docetaxel)

Females who are pregnant or lactating

Patients with peripheral neuropathy NCI-CTC grade 2 or greater

Patients who have received wide-field radiation, cytotoxic chemotherapy or hormonal therapy within 4 weeks of study entry; or mitomycin or nitrosoureas within 6 weeks of study entry

Patients who have had an investigational agent within 4 weeks of study entry

Patients receiving concurrent anticonvulsants known to induce P450 isoenzymes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2002-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Determine the Objective Response Rate | When all patients have completed treatment

SECONDARY OUTCOMES:
To determine time to disease progression | When all patients have completed treatment

CONTACTS AND LOCATIONS:
Locations (1):
- 5 Clinical Sites, 3 Cities, Russia